CLINICAL TRIAL: NCT00005732
Title: Develop and Implement Asthma Controlling Strategies (1)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4941
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-08

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
To develop and implement asthma controlling strategies for inner city and high risk populations.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a serious chronic disease affecting about 12 million Americans; about 3 million are children. The study was part of an initiative, "Developing and Implementing at the State and Local Level Educational Strategies and Interventions for Controlling Asthma in Inner City and High Risk Populations", released in February 1993 by the National Asthma Education Program of the Office of Prevention, Education and Control.

ELIGIBILITY:
No eligibility criteria

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Study Completion 1997-01